CLINICAL TRIAL: NCT05722392
Title: An IDEAL Phase 2a, Single-arm, Single-center, Prospective Study of Two-step Radical Prostatectomy in the Treatment of Low- to Intermediate-risk Prostate Cancer Concomitant With Severe Benign Prostatic Hyperplasia
Brief Title: Safety and Efficacy of Two-step Radical Prostatectomy
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Professor, Sun Yat-sen University
Other Study IDs: 2022-FXY-296
Record Dates: First submitted 2023-01-12; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Two-step Radical Prostatectomy: Two-step Radical Prostatectomy
  Interventions: Procedure: Two-step Radical Prostatectomy

INTERVENTIONS:
Procedure: Two-step Radical Prostatectomy — The first step is enucleation of the hyperplastic adenoma, and the second step is anterograde RP to residual gland

SUMMARY:
The goal of this observational study is to learn about the safety and efficacy of two-step radical prostatectomy in the treatment of low- to intermediate-risk prostate cancer patient with enlarged prostate and severe benign prostatic hyperplasia. The main question it aims to answer are: 1. Whether two-step prostatectomy is safe enough to decrease the surgical difficulty of these patients? 2. Whether the oncologic control is promising?

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as prostate cancer pathologically by prostate biopsy
2. Evaluated as localized prostate cancer by imaging studies
3. Prostate volume>70mL evaluated by transrectal ultrasonography or multi-parametric magnetic resonance imaging
4. Gleason score≤ 4+3=7
5. Preoperative PSA<20ng/mL
6. Estimated survival> 10 years；
7. Informed consent is obtained from the patient

Exclusion Criteria:

1. The patient has received other therapy including radical radiotherapy, transurethral resection of the prostate, cryoablation, HIFU, etc.
2. Any contraindication of surgery or anaesthesia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male with prostate cancer
Study Population: Low- to intermediate-risk localized prostate patient with enlarged prostate and severe benign prostatic hyperplasia
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2033-02-15 (Estimated); Study Completion 2033-02-15 (Estimated)

PRIMARY OUTCOMES:
Biochemical Recurrence-free Survival | 5 years
  Number of participants who are free of biochemical relapse after a specified duration of time. Biochemical recurrence is measured by PSA levels. Biochemical recurrence was defined as a measurable serum PSA concentration 0.2 ng/ml or greater.

SECONDARY OUTCOMES:
Surgical time | Intraoperative
  Defined as the time duration from the incision at the opening to the end of closing the incision
Estimated blood loss | Intraoperative
  Defined as all the blood loss counting during the surgery
Hospital stay | From date of surgery until the date of discharge, an average of 7 days
  Defined as the time duration between the first day after surgery to the day of discharge
Continence | 2 weeks, 1 months, 3 months, 6 months, 12 months after surgery
  Evaluated with the use of pad per day. Using no more than 1 pad per day is defined as complete continence
Lower urinary tract symptoms | 1 months, 3 months, 6 months, 12 months after surgery
  Evaluated with International Prostatic Symptom Score (IPSS). 1-7: Mild 8-19:Moderate 20-35: Severe
Erectile function | 6 months, 12 months and 24 months after surgery
  Evaluated with International Index of Erectile Function-5 (IIEF-5).The IIEF-5 score is the sum of the ordinal responses to the 5 items.
  22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction
Positive surgical margin rate | Through study completion, an average of 5 year
  Defined as the proportion of patients with positive surgical margin of the whole prostate and the margin between the hyperplastic adenoma and the residual gland evaluated by pathologists. The location of positive margin will be documented.
Complication | Through study completion, an average of 5 year
  All the complications which was evaluated relevant to the surgery will be documented and graded by Clavien-Dindo grade system.
Overall survival | From date of randomization until the date of date of death from any cause, assessed up to 60 months
  Number of participants who are alive after a specified duration of time
Cancer-specific survival | From date of randomization until the date of date of death from cancer, assessed up to 60 months
  Number of participants who are not dead due to prostate cancer after a specified duration of time

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No